CLINICAL TRIAL: NCT03871699
Title: The Effect of Ferric Carboximaltose on Intra-myocardial Iron Load Assessed by Cardiac Magnetic Resonance in Patients With Heart Failure With Reduced Ejection Fraction (HFREF).
Brief Title: Ferric Carboximaltose on Intra-myocardial Iron Load in Patients With Heart Failure
Acronym: IronHeart
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IronHeart
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Failure; Systolic Heart Failure; Heart Failure, Systolic
Keywords: Heart; Failure; Iron; Deficiency; Systolic; Reduced; Ejection
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Systolic Murmurs | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Iron Reposition (Experimental): The selected patients will receive 1g of ferric carboxymaltose applied intravenously after dilution in 100ml of crystalline solution. the infusion time will be around 15 minutes realized at the moinhos the vento infusion center.
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Ferric carboxymaltose — Administration of Ferric Carboxymaltose intravenously, one dose only.
  Other Names: Ferrinject

SUMMARY:
In general, anemia is associated with a greater presence of HF symptoms, worsening NYHA functional class, higher rate of hospitalization for heart failure, and reduced survival. However, it is unclear whether anemia is the cause of decreased survival or a marker for more advanced disease. Correction of iron deficiency in patients with New York Heart Association (NYHA) class II or III HF using intravenous iron (Ferinject®) improved "overall patient self-assessment" and NYHA functional class of 6-minute walk and health-related quality of life) in the FAIR-HF trial.

It is unknown if iron deficiency is correlated with intra-myocardial iron load as assessed by cardiac magnetic resonance (CMR) and if the treatment with intravenous iron has any impact on intra-myocardial iron load and left ventricular function.

The aim of the present study is to evaluate the effect of intravenous iron replacement on intra-myocardial iron deposits and the effect on left ventricular function.

Because it is a pilot study with few data in the literature, it is planned to use an initial sample of 20 patients.

We aim to evaluate the global ventricular function, the iron load by the T2 * method, the cardiac strain, the "Fiddle" and the "Fat water" of each patient by CMR. After this examination, patients will undergo intravenous infusion of 1g of Ferric Carboxymaltose (Ferinject®).

A comparative analysis of the ejection fraction values at the beginning and at the end of the study by CMR will be performed, in addition to a clinical reassessment.

The inclusion criteria will be: Patients older than 18 years, with iron deficiency and reduced ejection fraction defined as: serum ferritin <100 μg / L or with ferritin 100-299 μg / L with transferrin saturation <20 %; Hemoglobin <12g / dL in women and <13g / dL in men; Clinical stability in the last 3 months; Left ventricular ejection fraction (LVEF) <40% assessed by transthoracic echocardiography or CMR in the last 3 months. The exclusion criteria will be: patients with preserved ejection fraction (> 50%), pregnant women, refusal to participate in the present study, implantable pacemaker or implantable defibrillator incompatible with MRI, cerebral cerebral aneurysm clip and/or intracerebral or intraocular metal fragments, electronic cochlear implants, patients with claustrophobia, patients with clinical or hemodynamic instability and patients with indication for blood transfusion (Hb ≤ 7g / dL).

DETAILED DESCRIPTION:
Anemia (defined as a hemoglobin concentration below 13 g / dL in men and less than 12 g / dL in women) is a condition frequently associated with heart failure (HF), and its prevalence is estimated at around 4% to 50 %, depending on the study population and the adopted definition.

In general, anemia is associated with a greater presence of HF symptoms, worsening NYHA functional class, higher rate of hospitalization for heart failure, and reduced survival. However, it is unclear whether anemia is the cause of decreased survival or a marker for more advanced disease.

The etiology of anemia is multifactorial, including reduced sensitivity to erythropoietin receptors, presence of a hematopoiesis inhibitor and / or a defective iron supply for erythropoiesis. There is growing evidence that iron availability may be reduced absolutely due to decreased enteral iron absorption and / or occult hemorrhage, as well as in relative form, resulting from the dysregulation of iron homeostasis and accumulation of iron in cells of the reticuloendothelial system, characteristic of chronic disease anemia.

Recently, it has been suggested that iron deficiency itself may be an independent predictor of outcome in HF.

Correction of iron deficiency in patients with New York Heart Association (NYHA) class II or III HF using intravenous iron (Ferinject®) improved "overall patient self-assessment" and NYHA functional class of 6-minute walk and health-related quality of life) in the FAIR-HF trial. The treatment of patients with heart failure with mild to moderate anemia (hemoglobin levels from 9.0 to 12.0 g / dL) with the erythropoietin analogue, darbepoetin alfa was evaluated in the RED-HF trial (Reduction of Events with Darbepoetin Alfa in Heart Failure). No differences in the primary end point of death from any cause or hospitalization due to HF, or in the secondary outcome of cardiovascular death or time until the first hospitalization due to HF. The absence of darbepoetin was consistent across all subgroups. Of relevant, treatment with darbepoetin alfa led to an early increase (within one month) and sustained in the hemoglobin level throughout the study. These RED-HF trial results suggest that the level of hemoglobin, as well as other sub- stantial outcomes in HF, may be a prognostic marker, with decreased levels correlated with a worse prognosis, rather than a therapeutic target of HF.

A 2009 study tested the hypothesis of the association between anemia and HF severity, and the outcome could be explained by the emptying of iron stores, particularly at the myocardium level. This concept is based on previous experimental work showing that iron deficiency is associated with progressive left ventricular dysfunction and cardiac fibrosis.

Although serum ferritin is clinically used to estimate body iron stores, it reports approximately 1% of the total iron storage pool and its measurement can be confounded by a number of conditions, such as inflammation, abnormal liver function, and ascorbic acid deficiency. In contrast to serum ferritin, hepatic iron may serve as a better indicator of serum iron; however, it does not reflect myocardial iron. Cardiac iron overload and related toxicity may occur despite low hepatic iron concentrations.

Measurement of cardiac iron represented a major challenge to society. Endomyocardial biopsy is highly risky and potentially imprecise due to the small sample size and the heterogeneous deposition of cardiac iron. The introduction of cardiac magnetic resonance imaging (CMR) provided a reliable measure of tissue iron and revolutionized our understanding and management of iron-induced cardiomyopathy.

Iron, because is paramagnetic, can be quantified by Magnetic Resonance (MRI) in both the liver and the heart through a method called T2 * (T2 "star"). Myocardial iron deposition can be detected using myocardial T2 * and is the most important variable for predicting a need for treatment for ventricular dysfunction in the context of iron overload (eg, polytransfusion).

The clinically important iron load is defined as T2 * with values less than 20 ms, and is considered serious if it is less than 10 ms.

In 2016, a study in Spain evaluated patients with heart failure (with or without anemia) and their response to intravenous iron infusion. These patients, initially with mean T2* values of 39.5 msec, were followed by Cardiac Magnetic Resonance (CMR) before and after iron replacement with Ferric Carboxymaltose (Ferinject®) , obtaining at the end of the study, improvement in ventricular function and increase in the myocardial iron load (T2 * mean of 32 msec ).

The aim of the present study was to evaluate the correlation between intravenous iron replacement and increased intra-myocardial iron deposits and their effect on ventricular function.

In the CMR, the global ventricular function, the iron load by the "T2 * method", the cardiac "Strain" and the "Fat Water" of each patient will be analyzed. After this examination, patients will undergo intravenous 1g of Ferric Carboxymaltose (Ferinject®).

A comparative analysis of the ejection fraction values at the beginning and at the end of the study by CMR will be performed, in addition to a clinical reassessment, in which improvement of dyspnea and tiredness are expected.

There will be laboratory reassessment of ferritin and transferrin saturation to monitor treatment.

ELIGIBILITY:
Inclusion Criteria:

Left ventricular ejection fraction <40% assessed by transthoracic echocardiography or cardiac magnetic resonance with at least 3 months.

* Serum ferritin < 100µg/L or 100-299µg/L with transferrin saturation < 20%
* clinical stability during last 3 months

Exclusion Criteria:

* Use of intracardiac defibrillator or pacemaker.
* Severe to moderate valvar heart disease
* Clinical instability, acute coronary syndrome and cardiac surgery within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Absolut changes in left ventricular ejection fraction | 30 days
  Compare the left ventricular ejection fraction 30 days after receiving 1g of ferric carboxymaltose intravenously.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Beck da Silva, MD ScD, Principal Investigator — Hospital Moinhos de Vento; Luciano Giordani, MD, Study Director — Hospital Moinhos de Vento; Carisi A Polanczyk, MD ScD, Study Director — Hospital Moinhos de Vento; Paulo R Schvartzman, MD ScD, Study Director — Hospital Moinhos de Vento
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No